CLINICAL TRIAL: NCT03620734
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Study to Determine Interaction Between the Use of Feminizing Hormone Therapy and Antiretroviral Agents Concomitantly Among Transgender Women
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: iFACT
Record Dates: First submitted 2018-05-31; First posted 2018-08-08 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: PrEP and ART

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- GAHT and PrEP: HIV-negative TGW will have HIV testing using the 4th generation immunoassays/nucleic acid testing (NAT) in acute HIV testing algorithm currently used at the Thai Red Cross Anonymous Clinic at week 5, 8, and 15. Creatinine clearance will be performed at week 15.
- GAHT and ART: HIV-positive TGW on ART will have their plasma HIV RNA measured at the same day ART is initiated and at week 15 (12 weeks after ART provision). CD4 count will be measure at week 15.

SUMMARY:
Objective

1. To determine pharmacokinetic (PK) DDI between GAHT and ARVs used as PrEP and ART among TGW
2. To evaluate ARV adherence among TGW

DETAILED DESCRIPTION:
GAHT will be initiated on week 0. ARVs, either PrEP or ART, will be initiated on week 3. GAHT will then be withheld on week 5, and restart at week 8.

GAHT: Oral estradiol valerate 2 mg once daily and cyproterone acetate 25 mg once daily, which are the treatment of choice for GAHT in the TRC-ARC's Tangerine Community Health Center, will be provided to all participants.

PrEP and ART regimen: Generic fixed-dose combination of TDF 300 mg and FTC 200 mg will be used for PrEP and a generic fixed-dose combination of TDF 300 mg, FTC 200 mg and efavirenz 600 mg will be used for ART as recommended in the 2017 Thailand National Guidelines on HIV/AIDS Treatment and Prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Age 18-40 years old
3. Male-to-female transgender individual
4. PrEP/ART naïve
5. Body mass index 18.5-25 kg/m2
6. Calculated creatinine clearance (CrCl) ≥60 mL/min, as estimated by the Cockcroft- Gault equation
7. Alanine aminotransferase (ALT) ≤2.5 x ULN
8. Have signed the informed consent form

Exclusion Criteria:

1. Known history of allergy to hormonal or ARV component to be used in the study
2. Male-to-female transgender who underwent orchiectomy
3. Any of the following in HIV-infected participants

   * CD4 < 350 cells/mm3
   * History of psychiatric disorder that may be worsening by taking EFV
4. Previous use of injectable GAHT in the past 6 months
5. Current use of any of the following medication:

   * Anticonvulsant: Phenytoin, carbamazepine or phenobarbitol
   * Ergot-containing agents: dihydroergotamine, ergotamine or other ergot derivatives
   * Sedatives: Midazolam or triazolam
   * Herbs: Gingko biloba, St John's wort or milk thistle
   * Anti-infective agents: Erythromycin, clarithromycin, ketoconazole, itraconazole, rifampicin or rifabutin
6. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: transgender women (TGW)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Geometric mean (%CV) area under the plasma concentration time curve from 0 to 24 hours (AUC0-24) of estradiol | Measured at week 3 and week 5 of the study period
Geometric mean (%CV) area under the plasma concentration time curve from 0 to 24 hours (AUC0-24) of tenofovir | Measured at week 5 and week 8 of the study period
Geometric mean (%CV) maximum plasma concentration (Cmax) of estradiol | Measured at week 3 and week 5 of the study period
Geometric mean (%CV) maximum plasma concentration (Cmax) of tenofovir | Measured at week 5 and week 8 of the study period
Geometric mean (%CV) trough plasma concentration (C24) of estradiol | Measured at week 3 and week 5 of the study period
Geometric mean (%CV) trough plasma concentration (C24) of tenofovir | Measured at week 5 and week 8 of the study period
Geometric mean (%CV) half-life (t1/2) of estradiol | Measured at week 3 and week 5 of the study period
Geometric mean (%CV) half-life (t1/2) of tenofovir | Measured at week 5 and week 8 of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (1):
- The Thai Red Cross AIDS Research Centre, Ratchadamri, Bangkok, Thailand

REFERENCES:
- [Derived] Hiransuthikul A, Janamnuaysook R, Himmad K, Kerr SJ, Thammajaruk N, Pankam T, Phanjaroen K, Mills S, Vannakit R, Phanuphak P, Phanuphak N; iFACT Study Team. Drug-drug interactions between feminizing hormone therapy and pre-exposure prophylaxis among transgender women: the iFACT study. J Int AIDS Soc. 2019 Jul;22(7):e25338. doi: 10.1002/jia2.25338. PMID 31298497